CLINICAL TRIAL: NCT03091049
Title: Trans-radial Cardiac Catheterization Local Anesthesia: an Observational Study
Brief Title: RAOLA Observational: Local Anesthesia During Cardiac Catheterization
Status: Completed | Type: Observational
Sponsor: Hippocration General Hospital (Other)
Responsible Party: Principal Investigator, Dimitris Tousoulis, Professor of Cardiology, Hippocration General Hospital
Other Study IDs: RAOLA Observational
Record Dates: First submitted 2017-03-07; First posted 2017-03-27 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2018-02

CONDITIONS: Anesthesia, Local
Keywords: coronary; catheterization; transradial; anesthesia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EMLA anesthetic ointment (AO): In AO group a layer of 2.5 gr EMLA cream (standard adult dose) is applied to both wrists, 1 cm above the styloid process of the radius 30 minutes before the puncture, by an experienced cathlab nurse
- Local Skin Anesthetic Injection (LA): In LA group the radial artery is infiltrated with 1-2 mL of 2% lidocaine, using a 26 G needle, 0.5-1 cm proximal to the styloid process one minute before the puncture

SUMMARY:
An open label observational clinical study to compare the efficacy of EMLA cream (lidocaine 2.5% and prilocaine 2.5% in a ratio of 1:1 by weight) in comparison to the established local anesthesia (LA) protocol of lidocaine subcutaneous injection, in providing adequate peri-operative local anesthesia during transradial coronary angiography

DETAILED DESCRIPTION:
A total of 800 consecutive patients, who are referred for elective coronary angiography to 1st Cardiology Department cathlab, with the suspicion of coronary artery disease (CAD) will be enrolled in this study. Exclusion criteria are acute coronary syndrome, previous ipsilateral transradial approach, Raynaud's syndrome, abnormal renal function with or without need for hemodialysis, known history of sensitivity to local anesthetics, non-palpable radial pulse, abnormal Barbeau's test and patient's refusal. Baseline clinical, demographic and procedural data of the study population will be recorded.

The study will not involve any intervention but it will observe patients assigned to other EMLA cream or lidocaine injection for local anesthesia as part of their clinical routine treatment during transradial catherization.

Primary end-point: the perception of radial pain assessed during artery puncture and 30 minutes after sheath removal. Secondary end-point: The number of puncture attempts, the total time required before successful sheath insertion, and the occurrence of radial artery spasm will be also documented in each group Participants will be observed for 4 hours post angiography for development of local complications or side effects.

ELIGIBILITY:
Inclusion Criteria:

- patients, referred for elective diagnostic coronary angiography

Exclusion Criteria:

* acute coronary syndrome
* previous ipsilateral transradial approach
* Raynaud's syndrome
* abnormal renal function with or without need for hemodialysis
* known history of sensitivity to local anesthetics
* non-palpable radial pulse, abnormal Barbeau's test
* patient's refusal

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 800 consecutive patients, referred for elective coronary angiography In 1stCardiology Dpt Cath Lab with the suspicion of coronary artery disease (CAD) are enrolled in this study. All procedures will be undertaken by experienced and radial dedicated interventional cardiologists (i.e. more than 90% radial catheterizations). Exclusion criteria were acute coronary syndrome, previous ipsilateral transradial approach, Raynaud's syndrome, abnormal renal function with or without need for hemodialysis, known history of sensitivity to local anesthetics, non-palpable radial pulse, abnormal Barbeau's test and patient's refusal
Sampling Method: Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-10 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale of Pain Perception during sheath insertion | During artery puncture
  The primary end-point of the study is the perception of radial pain assessed during artery puncture

SECONDARY OUTCOMES:
Puncture efficiency | During radial artery catheterization
  The total time required for successful sheath insertion is documented in each group and constitutes the secondary end point of the study assessing puncture efficiency
Radial artery spasm | During radial artery catheterization
  The occurrence of radial artery spasm in each group during radial artery catheterization
Visual Analog Scale of Pain Perception 30 minutes after sheath removal | 30 minutes after sheath removal
  The primary end-point of the study is the perception of radial pain assessed 30 minutes after sheath removal

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Tousoulis, MD PhD, Study Director — 1st Cardiology Department - Athens Medical School
Locations (1):
- 1st Cardiology Department Hippokration Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No